CLINICAL TRIAL: NCT01040676
Title: The Use Of Automated Telephone Nutrition Support In Spanish-Speaking Latino Patients With Diabetes
Brief Title: Automated Telephone Nutrition Support
Acronym: ATNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121609ATNSUCSF
Record Dates: First submitted 2009-12-27; First posted 2009-12-29 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Telephone; Nutrition Support; Automated; Low English Proficiency; Hispanic; Latino
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients in this (the control group) will be eligible to receive the intervention (see "Intervention Group") after 12 weeks (essentially when the trial is over).
- Intervention Group (Experimental): Patients in the intervention group will receive automated telephone calls at regular intervals twice a week. The system will be programmed to call them at these intervals until contact. The ATNS system will solicit information from them in a culture specific manner, inquiring as to what foods they are eating each meal, each day, and each month. The ATNS system will then make proactive suggestions regarding low glycemic index foods, giving encouragement and feedback as appropriate.
  Interventions: Behavioral: Automated Telephone Nutrition Support

INTERVENTIONS:
Behavioral: Automated Telephone Nutrition Support — See Intervention Group description.
  Other Names: ATNS
  Arms: Intervention Group

SUMMARY:
The Automated Telephone Nutrition Support (ATNS) study investigates the effect of automated telephone nutrition support on diet and glycemic control among Spanish-speaking diabetics in Oakland.

DETAILED DESCRIPTION:
The Automated Telephone Nutrition Support (ATNS) study is a joint effort between the University of California at San Francisco, La Clinica de la Raza, and patients living with diabetes in Fruitvale (Oakland). Our goal is to see if motivated people with diabetes are able to get their blood sugar under better control by choosing a healthier diet. Since it's hard to eat a healthy diet, one of the ways we are trying to help is by calling people, having them record what they've eaten, and reminding them of the right foods to eat. The innovative part is using an automated telephone system to call them to have them record their dietary choices and giving them feedback immediately regarding what to modify as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Diabetic with A1c >8.5 for at least 1 year based on clinic records.
* Spanish-speaking (self-defined)

Exclusion Criteria:

* No telephone at home
* Planning to be out of town for longer than 2 weeks in the coming 12 weeks and thus unable to take part in follow up
* Pregnancy
* Insulin-dependent Diabetes
* Any evidence of end organ damage including chronic kidney disease requiring dialysis, congestive heart failure, or cirrhosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 weeks

SECONDARY OUTCOMES:
Weight | 12 weeks
Body Mass Index | 12 weeks
Blood Pressure | 12 weeks
Low Density Lipoprotein-calculated (LDL-c) | 12 weeks
C-reactive Protein | 12 weeks
Waist Circumference | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Gonzales, MD, MSPH, Principal Investigator — University of California, San Francisco
Locations (1):
- La Clinica de la Raza, Oakland, California, United States